CLINICAL TRIAL: NCT03089801
Title: Making Connections: Tablet-Enabled Video Telehealth to Enhance Veterans' Access and Care
Brief Title: Tablet-Enabled Video Telehealth to Enhance Veterans' Access and Care
Status: Completed | Type: Observational
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Donna Zulman, Principal Investigator, VA Palo Alto Health Care System
Other Study IDs: 1
Record Dates: First submitted 2017-03-09; First posted 2017-03-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2018-11

CONDITIONS: Chronic Disease, Mental Illness
Keywords: health care access; eHealth; telehealth
MeSH Terms: conditions — Chronic Disease; Mental Disorders | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tablet Recipients: Veteran patients who have received a VA-issued tablet for tablet-enabled video telehealth.
  Interventions: Other: Tablet-Enabled Video Telehealth
- Usual Care: Veteran patients who match tablet recipients based on sociodemographic/clinical characteristics but have not received a VA-issued tablet.

INTERVENTIONS:
Other: Tablet-Enabled Video Telehealth — Veterans referred for tablet-enabled video telehealth will receive a VA-issued tablet that can be used to communicate via video with health care providers (e.g., for chronic disease management, mental health treatment, palliative care).
  Other Names: eHealth
  Groups: Tablet Recipients

SUMMARY:
In order to enhance access to clinical and mental health services for Veterans who have geographic, clinical, or social barriers to in-person care, VA Offices of Connected Care and Rural Health began distributing 5,000 tablets to Veterans with access barriers in 2016. The objective of this Quality Improvement evaluation is to:

1. Understand characteristics of Veterans who received tablets, the frequency and ways in which they used the tablets, and the effects of tablet use on access to VA services.
2. Through a survey of Veterans, evaluate patient experiences using the tablets, and determine how tablets influenced patients' experiences with VA care, including their satisfaction, communication with providers, and access to needed services.
3. Identify implementation barriers and facilitators to tablet distribution and use through interviews with clinicians and staff in a purposive sample of VA facilities
4. Evaluate the effects of tablet use on chronic medical condition outcomes (e.g., hypertension, diabetes) and mental health treatment initiation and engagement (e.g., for depression, PTSD, and substance use).

DETAILED DESCRIPTION:
Background:

Telehealth is a cornerstone of enhanced access for Veterans and across a range of conditions is associated with improved disease control, quality of life, and patient satisfaction. Increasingly Veterans are able to monitor their chronic conditions and communicate with clinicians and care teams via tablets and other devices. However, this service is currently only available to Veterans with in-home Internet and video capability, or Veterans who are able to travel to a VA community based outpatient clinics to connect with providers at other facilities. In 2016, in order to address this access gap and disparity, VA launched an initiative to distribute tablets to Veterans who have clinical needs for remote care, and barriers to traditional in-person access.

Veterans who meet specific need-based (access, technology, and clinical) criteria may be issued one of two devices: Commercially available Off the Shelf (COTS) for basic connectivity or Healthcare Access Tablet (HAT) with a general exam camera and optional peripheral devices (i.e., stethoscope, BP monitor, pulse oximeter, thermometer, or weight scale). VA providers refer eligible patients for the devices using a consult template in VA's electronic health record. Care delivered via the tablet is indicated in the referral and may include one or more of the following: Home Based Primary Care, Palliative Care, Mental Health Intensive Case Management, Spinal Cord Injury, Mental Health Care, care for patients with marked mobility problems, care for patients with cognitive problems (these patients must have a caregiver who can assist with technology), home evaluations, and rehabilitation/prosthetics. Once the patient is issued the device, he or she will receive tablet services from trained teleproviders.

The VA began distributing tablets in the spring of 2016, with the plan of distributing 5,000 tablets over the following 1-2 years. Veteran eligibility criteria for tablets include the following: 1) Enrolled in VA Healthcare, 2) Does not own a device or does not have working broadband or cellular internet connection, 3) Physically and cognitively able to operate the technology (or has caregiver who can assist), 4) Barriers to access, such as a) distance or geography, b) transportation issues, c) homebound or difficulty leaving home, d) other (described by provider), and 5) Provider and patient give informed consent agreeing to utilize telehealth for care.

The tablet initiative and evaluation have been designated as Quality Improvement by VA's Office of Rural Health. The evaluation will include the following:

1. Tablet Recipient Characteristics, Use of Tablets, and Effects on Access. The investigators will first characterize Veterans who are issued and use the devices (e.g., age, sex, medical and mental health conditions, rural location/distance from VA). Investigators will describe the frequency of tablet use and the types of services that the Veteran receives (e.g., chronic disease management, mental health therapy, palliative care, home-based primary care). Investigators will analyze rates of in-person (outpatient, emergency care), telephone, and telehealth-based care before and after tablet distribution, and compare patterns to those observed in a cohort of comparable patients to assess whether tablets influence access and patterns of use.
2. Effects on Patient Experience. For patients receiving tablets beginning in March, 2017, the investigators will administer a survey at time of tablet receipt, and 3-6 months after that time, to examine changes in patients' satisfaction with VA care and their perceived access and communication, and to evaluate their experiences using the tablets. The survey will also assess patients' needs and risk factors (e.g., social support, health literacy), and how these factors impact patients' experiences with the tablets and VA care. If resources permit, the survey may be administered to a cohort of comparable patients who have not received tablets (to be determined as of March, 2017).
3. Implementation Evaluation. The implementation evaluation will be guided by the Consolidated Framework for Implementation Research (CFIR). The investigators will first administer an online survey to Facility Telehealth Coordinators (FTCs) at facilities that are distributing tablets. The survey will query FTCs about the tablet initiative, resources that facilitated implementation, and barriers that impeded implementation. The investigators will use survey responses to identify FTCs who represent a range of VA facilities (in terms of high vs. low tablet distribution rates). Follow-up interviews will be conducted by telephone. The investigators will transcribe and code the interviews using standard content analysis methods with the goal of understanding barriers and facilitators to tablet distribution within each of the CFIR domains.
4. Effects on Chronic Disease and Mental Health Outcomes. If resources are available in FY18, the investigators will evaluate how device distribution influences clinical outcomes for Veterans with common and high-risk conditions, such as hypertension, diabetes, and PTSD (conditions to be determined based on prevalence rates in the tablet recipient population). The investigators will compare measures of disease control (e.g., blood pressure readings, hemoglobin A1C levels) at 3 and 6 months after device shipment, and compare these levels to comparable patients from other facilities, using propensity scores to match patients on the basis of sociodemographic and clinical characteristics. The investigators will use similar methods to examine treatment initiation and engagement rates among patients with common mental health conditions, such as depression, PTSD, and substance use disorder.

The proposed project will be conducted with support from the eHealth Partnered Evaluation Initiative, a partnership between QUERI and Office of Connected Health that aims to evaluate the implementation of patient-provider technologies across VA, and understand their impacts on Veteran experience, perceived burdens and benefits to clinical teams, access to care, other care processes, and Veteran health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Veteran enrolled in a Veterans Affairs Health Care System, currently receiving care
* Must have a geographic, clinical, or social barrier that impedes access to in-person clinical and mental health services
* Veterans are referred for VA-issued tablets by their provider

Exclusion Criteria: All Veterans who receive VA-issued tablets will be included in the evaluation. Veterans may opt out of the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants are Veterans who have received care at a VA facility in the past year.
Sampling Method: Non-Probability Sample
Enrollment: 32186 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Utilization of VA Services | Up to 1 year after receipt of tablet
  Changes in patient use of VA services before/after receiving tablet

SECONDARY OUTCOMES:
Satisfaction with VA Care | Baseline and 6 months follow-up after receipt of tablet
  Survey-based measure of patient satisfaction with VA care
Access to VA Care | Baseline and 6 months follow-up after receipt of tablet
  Survey-based measure of patient perceived access to needed services
Communication with Providers | Baseline and 6 months follow-up after receipt of tablet
  Survey-based measure of patient perceived communication with providers
Evaluate feedback from the facilities that implement the tablet program | Beginning 1 year after initial implementation of the program during 2017-2018
  Assessment: Interview and survey questions on CFIR implementation constructs

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Zulman, MD, MS, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No